CLINICAL TRIAL: NCT06545058
Title: Safety Profile of Ropivacaine in Dorsal Penile Nerve Block for Male Circumcision: a Large Cohort Study in Children
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Ropopenile
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pain; Necrosis
Keywords: Circumcision; Pain; Necrosis; Ropivacaine
MeSH Terms: conditions — Pain; Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: All male children aged up to 16 years, who underwent a circumcision at UZ Brussel, between 1 January 2000 and 31 December 2021
  Interventions: Procedure: Penile block

INTERVENTIONS:
Procedure: Penile block — Penile block with local anesthetics

SUMMARY:
Dorsal penile nerve block (DPNB) according to Dalens' technique by using local anesthetics (LAs) is a fundamental part of a multimodal analgesic approach following circumcision. Ropivacaine has a favorable cardiovascular and neurological toxicity profile. However, its application in DPNB is limited because of the theoretical concerns about its vasoconstrictive properties and the potential risks of ischemia of the glans. The aim is to evaluate the incidence of necrosis of the glans penis and the safety profile of ropivacaine following its use in the DPNB in a large pediatric population.

DETAILED DESCRIPTION:
Circumcision is one of the most practiced surgical procedures in childhood causing significant postoperative pain in the infant. Perioperative and postoperative pain management at this age ideally should be managed by a combination of general anesthesia with regional anesthesia techniques such as caudal block, dorsal penile nerve block or subcutaneous ring block of the penis.

The dorsal nerves of the penis can be anesthetized at the level of the penile root through different approaches. Kirya and Wertgmann described for the first time dorsal penile nerve block. Since then, many studies have been realized and have been showed its benefits and safety in the clinical use.

Ring Blok is also known for its safety and low incidence of complications and has been used primarily for postoperative pain management in circumcision. This block is easy to perform but it has been identified that it has a greater failure compared to the dorsal penile block. In the study of Holder who compares dorsal penile block and ring block, most of the children who has had a ring block also received opioids postoperatively.

Implementation of local or regional anesthesia techniques is inevitably associated with risks and complications. For DPNB, this is estimated around 0.18%. Those complications may include urethral injuries, accidental injection of an incorrect drug or drug dose, accidental intravascular injection of local anesthetics, ischial osteomyelitis, hematoma, and ischemia and necrosis of the glans penis. The dorsal nerves of the penis also lies close to de corpora cavernosa and the Buck's fascia. Given the rich vascularized features of these structure, DNPB may increase the risk of intravascular injection, systemic absorption of local anesthetics or hematoma.

Ischemia or even necrosis of the glans due to the placement of a penile block is a very rare complication that is not seen in the daily practice. Endothelial injury and necrosis is a serious complication that can be caused due to vascular compression because of the mass effect of anesthetic solution or hematoma, perforation of a vein or artery, excessive cauterization, a very tight suture, veno/vasospasm at the glans; secondary to surgery or the dorsal penile nerve block.

Ischemia or necrosis may also be due to the vasoconstrictive effect of local anesthetics, especially if they contain epinephrine.

Cases of ischemia of the glans have been described after the application of the dorsal penile nerve block, this was related to anesthetics that contained epinephrine or another type of vasoconstrictor agent.

Ropivacaine is a local anesthetic drug with a remarkable safe cardiologic and neurologic toxicity profile specially in children. Its administration for dorsal penile nerve block (DPNB) in male penile surgeries, however, has been discouraged because of the fear to cause necrosis of the glans due to its vasoconstrictor properties. In Universitair Ziekenhuis Brussel, we use ropivacaine for this purpose for more than 20 years now with seemingly no significant complications. We want to evaluate the safety of our practice that is associated with the use of ropivacaine in DPNB in the pediatric population, as well as the incidence and type of potential complications. The impact may be important because there are no studies that verify the safety of this local anesthetic for those type of procedures. This cohort study could eventually also serve as quality improvement.

Ropivacaine is a local anesthetic amide-type that has been shown to have vascular biphasic effects, with vasoconstrictive qualities. These properties have been verified in Dahl's study. Where they identified a decrease in epidural blood flow of 37%, compared to the increase in blood flow that they identified after the administration of bupivacaine.

The vasoconstrictive qualities have been related with low ropivacaine concentrations like 0.063% and 0.125%. At higher concentrations like 0.75% has been showed just a little decrease in blood flow comparing with saline. There are currently no other studies in the literature that indicate the risk of using ropivacaine in children for Dorsal Penile Nerve Block (DPNB).

ELIGIBILITY:
Inclusion Criteria:

* All male children aged up to 16 years
* All circumcision made at UZ Brussel
* All revision of circumcision made at UZ Brussel
* All procedures between 1 January 2000 and 31 December 2021
* All type ASA
* Penile Block performed by anesthesiologist
* All Penile Block performed with local anesthetics at diverse concentrations

Exclusion Criteria:

* Canceled procedure
* Missing anesthetic records
* Children who received caudal block by anesthesiologist in charge
* Children who received local infiltration of local anesthetics by the surgeon

Max Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: All children aged up to 16 years who underwent a circumcision at UZ Brussel, between 1 January 2000 and 31 December 2021
Sampling Method: Non-Probability Sample
Enrollment: 2086 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Incidence of necrosis of the glans penis | During time of surgery
  To evaluate the incidence of necrosis of the glans penis following the use of ropivacaine in the Dorsal penile nerve block in a large pediatric population.
Safety profile of Ropivacaine | During time of surgery
  To evaluate the safety profile of ropivacaine following its use in the Dorsal penile nerve block in a large pediatric population.

REFERENCES:
- [Background] Teunkens A, Van de Velde M, Vermeulen K, Van Loon P, Bogaert G, Fieuws S, Rex S. Dorsal penile nerve block for circumcision in pediatric patients: A prospective, observer-blinded, randomized controlled clinical trial for the comparison of ultrasound-guided vs landmark technique. Paediatr Anaesth. 2018 Aug;28(8):703-709. doi: 10.1111/pan.13429. Epub 2018 Jul 23. PMID 30035357
- [Background] Sfez M, Le Mapihan Y, Mazoit X, Dreux-Boucard H. Local anesthetic serum concentrations after penile nerve block in children. Anesth Analg. 1990 Oct;71(4):423-6. doi: 10.1213/00000539-199010000-00019. No abstract available. PMID 2205131
- [Background] Garrido-Abad P, Suarez-Fonseca C. Glans ischemia after circumcision and dorsal penile nerve block: Case report and review of the literature. Urol Ann. 2015 Oct-Dec;7(4):541-3. doi: 10.4103/0974-7796.164862. PMID 26692685
- [Background] Irwin MG, Cheng W. Comparison of subcutaneous ring block of the penis with caudal epidural block for post-circumcision analgesia in children. Anaesth Intensive Care. 1996 Jun;24(3):365-7. doi: 10.1177/0310057X9602400311. PMID 8805893
- [Background] Sara CA, Lowry CJ. A complication of circumcision and dorsal nerve block of the penis. Anaesth Intensive Care. 1985 Feb;13(1):79-82. doi: 10.1177/0310057X8501300111. No abstract available. PMID 3977067
- [Background] Jansson JR. Vasoactivity of ropivacaine. Reg Anesth Pain Med. 2008 Jan-Feb;33(1):90-1; author reply 91-2. doi: 10.1016/j.rapm.2007.08.011. No abstract available. PMID 18155065
- [Background] Doye E, Desgranges FP, Stamm D, de Queiroz M, Valla FV, Javouhey E. [Severe local anesthetic intoxication in an infant undergoing circumcision]. Arch Pediatr. 2015 Mar;22(3):303-5. doi: 10.1016/j.arcped.2014.10.023. Epub 2014 Nov 15. French. PMID 25482996
- [Background] Burke D, Joypaul V, Thomson MF. Circumcision supplemented by dorsal penile nerve block with 0.75% ropivacaine: a complication. Reg Anesth Pain Med. 2000 Jul-Aug;25(4):424-7. doi: 10.1053/rapm.2000.7594. PMID 10925943
- [Background] Wang X, Dong C, Beekoo D, Qian X, Li J, Shang-Guan WN, Jiang X. Dorsal Penile Nerve Block via Perineal Approach, an Alternative to a Caudal Block for Pediatric Circumcision: A Randomized Controlled Trial. Biomed Res Int. 2019 Mar 27;2019:6875756. doi: 10.1155/2019/6875756. eCollection 2019. PMID 31032356
- [Background] Mittino I, Sangalli M, Fabbri F, Sozzi F, Ghezzi M, Zanni G, Cestari A. Ischemia of the glans 24 hours after circumcision: A case report and therapeutic solution. Urologia. 2018 Nov;85(4):174-176. doi: 10.1177/0391560318761288. Epub 2018 Mar 26. PMID 30426879
- [Background] Lander J, Brady-Fryer B, Metcalfe JB, Nazarali S, Muttitt S. Comparison of ring block, dorsal penile nerve block, and topical anesthesia for neonatal circumcision: a randomized controlled trial. JAMA. 1997 Dec 24-31;278(24):2157-62. PMID 9417009
- [Background] Holder KJ, Peutrell JM, Weir PM. Regional anaesthesia for circumcision. Subcutaneous ring block of the penis and subpubic penile block compared. Eur J Anaesthesiol. 1997 Sep;14(5):495-8. doi: 10.1046/j.1365-2346.1997.00180.x. PMID 9303286
- [Background] Dahl JB, Simonsen L, Mogensen T, Henriksen JH, Kehlet H. The effect of 0.5% ropivacaine on epidural blood flow. Acta Anaesthesiol Scand. 1990 May;34(4):308-10. doi: 10.1111/j.1399-6576.1990.tb03092.x. PMID 2343734
- [Background] Najafi N, Veyckemans F, Du Maine C, van de Velde A, de Backer A, Vanderlinden K, Poelaert J. Systemic Toxicity Following the Use of 1% Ropivacaine for Pediatric Penile Nerve Block. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):549-50. doi: 10.1097/AAP.0000000000000415. No abstract available. PMID 27315186